CLINICAL TRIAL: NCT00381693
Title: Phase II Study of Azacitidine in Myelofibrosis
Brief Title: Azacitidine in Treating Patients With Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of accrual and trial has demonstrated too little clinical benefit
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Ruben A. Mesa, Mayo Clinic Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000503972; P30CA015083 (NIH); MC058D (Other: Mayo Clinic Cancer Center); 05-004297 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Myeloproliferative Disorders; Secondary Myelofibrosis
Keywords: primary myelofibrosis; polycythemia vera; essential thrombocythemia; secondary myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Polycythemia Vera; Thrombocythemia, Essential | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: azacitidine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of abnormal cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well azacitidine works in treating patients with myelofibrosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of azacitidine in patients with myelofibrosis (MF) with myeloid metaplasia.
* Evaluate the safety of azacitidine in these patients. Secondary
* Evaluate pertinent biologic characteristics of MF before and during therapy with azacitidine.
* Assess the effects of study treatment on constitutional symptoms in these patients.
* Estimate time to event distributions for overall survival and progression. OUTLINE: Patients receive azacitidine subcutaneously once daily on days 1-5. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed myelofibrosis with myeloid metaplasia (MMM), including any of the following subtypes:

  * Agnogenic myeloid metaplasia
  * Post-polycythemic myeloid metaplasia
  * Post-thrombocythemic myeloid metaplasia
* Evaluable and symptomatic disease, defined as 1 of the following:

  * Anemia (hemoglobin < 10 g/dL or erythrocyte transfusion-dependent, requiring 1 transfusion ≤ 8 weeks)
  * Treatment required* for symptomatic palpable splenomegaly (palpable hepatomegaly is acceptable if previously splenectomized) NOTE: *Subjective but painful enough to mandate intervention
* Absence of t(9;22) by fluorescent in situ hybridization (FISH) or standard cytogenetics (by peripheral blood or marrow)

  - Previous demonstration of a lack of this translocation (at any point) is sufficient
* No advanced malignant hepatic tumors

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 50,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 2.0 mg/dL OR direct bilirubin ≤ 2.0 mg/dL if total bilirubin elevated (unless attributed to underlying disease)
* AST and ALT ≤ 2 times upper limit of normal (unless clinically attributed to hepatic extramedullary hematopoiesis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No baseline peripheral or autonomic neuropathy ≥ grade 2
* No condition, including the presence of laboratory abnormalities, that would preclude study compliance
* No hypersensitivity to mannitol or azacitidine
* Not incarcerated in a municipality (i.e., county, state, or federal prison)

PRIOR CONCURRENT THERAPY:

* At least 14 days since prior chemotherapy, including interferon alfa, anagrelide, or other myelosuppressive agents
* At least 14 days since prior systemic corticosteroids
* At least 14 days since prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A. Mesa, MD, Study Chair — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten patients were recruited from August 2006 to December 2007 at Mayo Clinic. This trial was permanently closed in December 2007 due to lack of accrual and it demonstrated too little clinical benefit.
Groups:
- Azacitidine: Azacitidine 75 mg/m^2 subcutaneously
Period: Overall Study
Arm/Group | Azacitidine
Started | 10
Completed | 2
Not Completed | 8
Not completed — Death | 1
Not completed — Adverse Event | 4
Not completed — Patient Choice | 1
Not completed — Progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Azacitidine
Number analyzed (Participants) | 10
Age Continuous [Median (Full Range); unit: years] | 72 [57 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10
Disease [Number; unit: participants]
  Primary Myelofibrosis | 8
  Post-polycythemia Vera Myelofibrosis | 1
  Post-essential Thrombocythemia Myelofibrosis | 1
Lilie Score at Diagnosis (Myelofibrosis only) [Number; unit: participants] — A scoring system reported by Dupriez et al, which was constructed with the two adverse prognostic factors, namely Hb < 10 g/dL and WBC < 4 or > 30 x 10(9)/L, used to separate patients in three groups with low (0 factor), intermediate (1 factor), and high (2 factors) risks, associated with a median survival of 93, 26, and 13 months, respectively.
  participants
    0 (Low Risk) | 2
    1 (Intermediate Risk) | 5
    2 (High Risk) | 3
Red Cell Transfusion-dependent [Number; unit: participants]
  Yes | 7
  No | 3
Prior Thrombosis or Hemorrhage [Number; unit: participants]
  Yes | 0
  No | 10
Prior Therapy for Myelofibrosis [Number; unit: participants]
  Yes | 7
  No | 3

OUTCOME MEASURES:

1. Primary Outcome: Patients With Confirmed Response (Complete Remission or Partial Remission on 2 Consecutive Evaluation at Least 4 Weeks Apart) During the First 4 Months of Treatment
Description: Response Definitions:
  * Completion Remission (CR):complete resolution of disease-related symptoms, ultrasound-documented resolution of hepastosplenomegaly, normalization of the peripheral blood count, white cell differential, and smear, normalization of bone marrow histology including disappearance of fibrosis and osteosclerosis. Residual cytogenetic abnormalities are allowed.
  * Partial Remission (PR): a major response in any baseline applicable criteria (except constitutional symptoms) without progression in any other category.
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 10
participants | 0

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from registration to death due to any cause or time from registration to 3 years after registration if patient is still alive.
Time Frame: From date of registration until death or 3 years after registration if patient is still alive
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine
Number analyzed (Participants) | 10
months | 16.9 [10.7 to 21.2]

3. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the time from registration to progression of disease. Those who die without documentation of disease progression will be considered to have had disease progression at the time of their death unless documented evidence clearly indicates no progression has occured.
Time Frame: up to 3 years
Population: Only 2 out of 10 patients had disease progression. One patient progressed at 0.5 months after registration and one patient progressed at 2.8 months after registration. Thus, median of time to progression and upper limit of 95% confidence interval are not attainable.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Treatment Related Adverse Events
Description: Adverse events (AE) that are classified as either possibly, probably, or definitely related to study treatment according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE version 3.0). The maximum grade for each type of AE will be recorded for each patient. Grade refers to the severity of the AE.
  Grade 1: Mild AE, Grade 2: Moderate AE, Grade 3: Severe AE, Grade 4: Life-threatening or disabling AE, Grade 5: Death related AE
Time Frame: Every 4 weeks during treatment
Measure: Number; unit: Participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 10
Participants
  Grade 1-2 Hematologic | 1
  Grade 3-4 Hematologic | 8
  Grade 1-2 Non-hematologic | 23
  Grade 3-4 Non-hematologic | 0

ADVERSE EVENTS:
Arm/Group | Azacitidine
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 2 (3)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine (N=10)
Anemia (Blood and lymphatic system disorders) | 5 (8)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 6 (8)
Vomiting (Gastrointestinal disorders) | 5 (6)
Edema Limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (24)
Leukopenia (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 5 (18)
Platelet count decreased (Investigations) | 7 (24)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes